CLINICAL TRIAL: NCT03182088
Title: Norepinephrine Infusion for Prevention of Post-spinal Hypotension During Cesarean Delivery: A Randomized Controlled Dose Finding Trial.
Brief Title: Norepinephrine Infusion Different Doses in Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-49-2017
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Bupivacaine; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0.025 mcg /Kg/min group (Experimental): The patients will receive spinal anesthesia through 10 mg Bupivacaine, then start norepinephrine bitartrate infusion (0.05 mcg/Kg/min) equivalent to norepinephrine infusion (0.025 mcg/Kg/min).
  Interventions: Drug: norepinephrine infusion (0.025 mcg/Kg/min); Drug: Bupivacaine
- 0.050 mcg/Kg/min group (Experimental): The patients will receive spinal anesthesia through 10 mg Bupivacaine, then start norepinephrine bitartrate infusion (0.1 mcg/Kg/min) equivalent to norepinephrine infusion (0.050 mcg/Kg/min).
  Interventions: Drug: norepinephrine infusion (0.050 mcg/Kg/min); Drug: Bupivacaine
- 0.075 mcg/Kg/min group (Experimental): The patients will receive spinal anesthesia through 10 mg Bupivacaine, then start norepinephrine bitartrate infusion (0.15 mcg/Kg/min) equivalent to norepinephrine infusion (0.075 mcg/Kg/min)
  Interventions: Drug: norepinephrine infusion (0.075 mcg/Kg/min); Drug: Bupivacaine

INTERVENTIONS:
Drug: norepinephrine infusion (0.025 mcg/Kg/min) — The patients will receive a bolus of 5 mcg norepinephrine followed by norepinephrine bitartrate infusion of (0.05 mcg/Kg/min) equivalent to norepinephrine base of (0.025 mcg/Kg/min)
  Other Names: noradrenaline infusion
  Arms: 0.025 mcg /Kg/min group
Drug: norepinephrine infusion (0.050 mcg/Kg/min) — The patients will receive a bolus of 5 mcg norepinephrine followed by norepinephrine infusion of (0.1 mcg/Kg/min) equivalent to norepinephrine base of (0.050 mcg/Kg/min)
  Other Names: noradrenaline infusion
  Arms: 0.050 mcg/Kg/min group
Drug: norepinephrine infusion (0.075 mcg/Kg/min) — The patients will receive a bolus of 5 mcg norepinephrine followed by norepinephrine infusion of (0.15 mcg/Kg/min) equivalent to norepinephrine base of (0.075 mcg/Kg/min).
  Other Names: noradrenaline infusion
  Arms: 0.075 mcg/Kg/min group
Drug: Bupivacaine — The patient will receive spinal anesthesia using Bupivacaine (10 mg).
  Other Names: spinal anesthesia; Heavy marcaine

SUMMARY:
three doses (0.025 mcg/Kg/min, 0.050 mcg/Kg/min, and 0.075 mcg/Kg/min) of norepinephrine will be compared for prophylaxis against Post-spinal anesthesia hypotension during Cesarean delivery.

DETAILED DESCRIPTION:
Maternal hypotension is a common complication after spinal anesthesia for cesarean delivery (CD). Using vasopressors have been considered a gold standard for prevention of post-spinal hypotension (PSH) during CD.

Norepinephrine (NE) is a potent vasopressor characterized by both α adrenergic agonist activity in addition to a weak β adrenergic agonist activity; thus, NE is considered a vasopressor with minimal cardiac depressant effect; these pharmacological properties would make NE an attractive alternative to phenylephrine and ephedrine (the most commonly used vasopressors in obstetric anesthesia).

Norepinephrine has been recently introduced as a prophylactic vasopressor during CD with promising results; However, the optimum dose for efficient prophylaxis with the least side effects is not known.

In this study, three doses (0.025, 0.050, 0.075 mcg/Kg/min) of norepinephrine will be compared for prophylaxis against PSH during CD.

ELIGIBILITY:
Inclusion Criteria:

* full term
* singleton
* pregnant women
* scheduled for elective cesarean delivery

Exclusion Criteria:

* cardiac morbidities
* hypertensive disorders of pregnancy
* peripartum bleeding
* baseline systolic blood pressure (SBP) < 100 mmHg
* body mass index > 35 will be excluded from the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 284 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-12-25 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
postspinal hypotension | 30 minutes after spinal anesthesia
  The number of patients who develop hypotension (defined as decreased SBP less than 80% of the baseline reading during the period from intrathecal injection till delivery of the fetus) after spinal block divided by the total number in the group

SECONDARY OUTCOMES:
severe postspinal hypotension | 30 minutes after spinal anesthesia
  The number of patients who develop hypotension (defined as decreased SBP less than 60% of the baseline reading during the period from intrathecal injection till delivery of the fetus) after spinal block divided by the total number in the group
Post-delivery hypotension | 10 minutes after delivery
  number of patients who develop hypotension (defined as decreased SBP less than 80% of the baseline reading after delivery of the fetus and starting oxytocin infusion)
systolic blood pressure | 60 minutes after spinal block
  systolic blood pressure measured in mmHg
diastolic blood pressure | 60 minutes after spinal block
  diastolic blood pressure measured in mmHg
heart rate | 60 minutes after spinal block
  heart rate measured in beats per minute
intraoperative hypertension | 60 minutes after spinal block
  number of patients who develop intraoperive hypertension (defined as increased systolic blood pressure by more than 20% of the baseline reading) divided by the total number of patients in the group
incidence of nausea and vomiting | 60 minutes after spinal block
  number of patients who develop nausea and vomiting divided by the total number of patients in the group
ephedrine consumption | 60 minutes after spinal block
  total amount of ephedrine consumed during the operation (measured in milligrams)
Atropine consumption | 60 minutes after spinal block
  total amount of atropine consumed during the operation (measured in milligrams)
APGAR score | 1 minute after delivery
  APGAR score for detection of the well being of the fetus
APGAR score | 10 minutes after delivery
  APGAR score for detection of the well being of the fetus

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mukhtar, Professor, Study Director — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No